CLINICAL TRIAL: NCT06960655
Title: Improving Lipid Optimization Quality and Treatment Options in ASCVD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Benjamin M. Scirica, MD, Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000910
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypercholesterolemia; ASCVD
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Provider Notification Strategy Procedures:
  The provider notification recommendations are based on current professional society guidelines with FDA-approved therapeutics. Providers may follow, modify, or reject those recommendations as they deem clinically most appropriate.
  Remote Pharmacist-driven Medication Management Strategy Procedures:
  Treatment recommendations in this program are based on current professional society guidelines with FDA-approved therapeutics. This program is based on a statutory-defined Collaborative Drug Therapy Management agreement approved by the BWH Pharmacy and Therapeutic Committee to initiate and titrate lipid-lowering medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EHR-Based Provider Notification for Lipid Optimization (Active Comparator)
  Interventions: Behavioral: Best-Practice Alert
- Remote Pharmacist-Driven Medication Management Program (Active Comparator)
  Interventions: Behavioral: Referral to Pharmacist-Driven Medication Management Program

INTERVENTIONS:
Behavioral: Referral to Pharmacist-Driven Medication Management Program — Medication initiations and titrations are based on an established drug-treatment algorithm that utilizes a statutory-defined Collaborative Drug Therapy Management Agreement (CDTM) approved by the BWH Pharmacy and Therapeutic Committee to initiate and titrate lipid-lowering medications. Scenarios outside the prescribed medication algorithm are routed to the supervising physician, and changes are signed off by a pharmacist and communicated to the patient and care team by a patient navigator under the supervision of physicians. After each change in medication, re-assessment and lab monitoring are collected in an iterative process until targets are achieved. Details of the programs can be found in the references.
  Arms: Remote Pharmacist-Driven Medication Management Program
Behavioral: Best-Practice Alert — This strategy will employ automated, asynchronous, best-practice alerts (BPAs). Provider notifications via electronic health records (EHRs) are clinical tools designed to improve adherence to evidence-based guidelines by providing real-time alerts that have been widely implemented across healthcare systems to enhance patient safety, reduce clinical inertia, and standardize care delivery. However, their effectiveness depends on factors such as alert fatigue, provider engagement, and integration into existing workflows. BPAs are one of the most common types of automated EHR-based provider notifications.
  Arms: EHR-Based Provider Notification for Lipid Optimization

SUMMARY:
The goal of this project is to study different approaches to improve the utilization of guideline directed medicines to lower cholesterol in patients with or at high risk of atherosclerosis (cholesterol buildup in the arteries).

DETAILED DESCRIPTION:
This project will include approximately 300 patients who, based on current guidelines, would benefit from optimized lipid management. The project is testing the most effective methods to notify providers and patients and inform them that their patients may benefit from further lipid optimization. It will utilize systematic allocation at the provider level in which clinicians are assigned to either the direct Provider Notification Strategy or the Pharmacist-Driven Medication Management Strategy, ensuring that all patients continue to receive guideline-based care while eliminating the risk of treatment selection bias. Approximately 100 providers to ensure a sufficient number of patients are included.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old and <=95 years old
* Established Atherosclerotic Cardiovascular Disease
* Diabetes
* Possible Familial Hypercholesterolemia (FH)
* High-Risk Primary Prevention

Exclusion Criteria:

* No PCP, cardiologist, endocrinologist, or nephrologist at MGB
* ESRD on dialysis
* Enrolled in a hospice program
* Advanced dementia

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Achieving Goal LDL-C | 6 months after notification
  % of participants who achieve LDL-c goal (<100 mg/dL for high-risk primary prevention, <70 mg/dL for patients with established ASCVD)

SECONDARY OUTCOMES:
Intensification lipid-lowering therapy | 12 months after notification
  % of participants who receive any intensification lipid-lowering therapy
Achieving Goal LDL-C | 12 months after notification
  % of participants who achieve LDL-c goal (<100 mg/dL for high-risk primary prevention, <70 mg/dL for patients with established ASCVD)
LDL- c reduction | 12 months after notification
  Total and average LDL-c reduction compared to baseline
Lipid testing and prescriptions | 12 months after notification
  Number of lipid-related lab testing or prescriptions for lipid-lowering therapy (by provider or remote disease management program; process related outcomes (responses to provider notifications)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Scirica, M.D., MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No